CLINICAL TRIAL: NCT00417755
Title: Effect of Invasive and Non Invasive Mechanical Ventilation on the Nutritional Status of COPD Elderly Patients
Brief Title: Effect of Invasive and Non Invasive Mechanical Ventilation on Feeding Delivery in COPD Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Other Study IDs: 4108
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2006-12

CONDITIONS: COPD; Mechanical Ventilation
Keywords: Nutritional intake; Mechanical ventilation; Enteral feeding
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
COPD patients requiring ventilation may benefit from invasive or non invasive ventilation. Non invasive ventilation is often incompatible with oral or enteral feding, due to gastric dilatation and full mask therapy. At the other hand, invasive ventilation is associated with incomplete enteral feeding and nutrition requirements are not reached. The aim of the study was to compare the feeding delivery of COPD patients receiving invasive or non invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients requiring mechanical ventilation (invasive and non invasive)

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-01; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, MD, Principal Investigator — Rabin Medical Center, Beilison Hospital, Israel